CLINICAL TRIAL: NCT02830763
Title: Clinical Study on the Safety and Efficacy of Medium-chain Fatty Acid Capsules (CNT-02) for Primary Triglyceride Deposit Cardiomyovasculopathy (TGCV) and Neutral Lipid Storage Disease With Myopathy (NLSD-M)
Brief Title: Clinical Study on the Safety of CNT-02 for TGCV and NLSD-M
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICVD1527; UMIN000023043 (Other: UMIN-CTR)
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Primary Triglyceride Deposit Cardiomyovasculopathy (TGCV); Neutral Lipid Storage Disease With Myopathy (NLSD-M)
Keywords: neutral lipid storage disease; CNT-02; primary triglyceride deposit cardiomyovasculopathy (TGCV); neutral lipid storage disease with myopathy (NLSD-M)
MeSH Terms: conditions — Neutral Lipid Storage Disease with Myopathy; Chanarin-Dorfman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medium-chain Fatty Acid (CNT-02) (Experimental)
  Interventions: Dietary Supplement: CNT-02

INTERVENTIONS:
Dietary Supplement: CNT-02 — Each subject will take 2.0g of the investigational product orally 3 times a day after every meal. Unless an apparent worsening of symptoms or unacceptable adverse event occurs, the subject will continue to take the investigational product for up to 6 months.

SUMMARY:
This study is planning to evaluate the safety and clinical efficacy of medium-chain fatty acid capsules (food-grade CNT-02) in subjects with primary triglyceride deposit cardiomyovasculopathy (TGCV) and neutral lipid storage disease with myopathy (NLSD-M) associated with adipose triglyceride lipase (ATGL) genetic defects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients for whom ATGL gene deletion has been previously confirmed.
2. Patients who can take the investigational product orally.
3. Male and female who are at least 20 years old at the time of consent.
4. Patients who gave written informed consent.

Exclusion Criteria:

1. Patients with diabetic ketoacidosis.
2. Patients with the possibility of diabetic ketoacidosis (patients with poorly controlled diabetes mellitus [HbA1c>8.4%, NGSP])
3. Patients with terminal malignancy.
4. Pregnant or lactating women.
5. Patients who do not consent to using contraception while participating in this study.
6. Patients allergic to MCT oil.
7. Patients participating in other clinical trial.
8. Otherwise, patients determined to be ineligible for this study by the investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
The maximum walking distance in a 6-minute walk test at 3 months | 3 months
  Measuring maximum walking distance of 6-minute walk test. Calculating variation of those measured values from baseline to 3 months.
The maximum walking distance in a 6-minute walk test at 6 months | 6 months
  Measuring maximum walking distance of 6-minute walk test . Calculating variation of those measured values from baseline to 6 months.

SECONDARY OUTCOMES:
MRC sum score in manual muscle testing (MMT) at 3 months | 3 months
  Evaluating muscle strength by manual muscle test used MRC score. Assessing change from baseline to 3 months.
MRC sum score in manual muscle testing (MMT) at 6 months | 6 months
  Evaluating muscle strength by manual muscle test used MRC score. Assessing change from baseline to 6 months.
Fractions of lung volume such as % vital capacity, measured by spirometer at 3 months | 3 months
  Evaluating the respiratory functions by % Vital capacity measured by spirometer. Assessing change from baseline to 3 months.
Fractions of lung volume such as % vital capacity, measured by spirometer at 6 months | 6 months
  Evaluating the respiratory functions by % Vital capacity measured by spirometer. Assessing change from baseline to 6 months.
The amount of fat measured by computed tomography (CT) of the skeletal muscle (fat deposition) at 3 months | 3 months
  Evaluating fat deposition in the skeletal muscle by CT. Assessing change from baseline to 3 months.
The amount of fat measured by computed tomography (CT) of the skeletal muscle (fat deposition) at 6 months | 6 months
  Evaluating fat deposition in the skeletal muscle by CT. Assessing change from baseline to 6 months.
Parameters of cardiac function, such as the left ventricular ejection fraction by echocardiography at 3 months | 3 months
  Evaluating cardiac function using Left ventricular ejection fraction etc. by echocardiography. Assessing change from baseline to 3 months.
Parameters of cardiac function, such as the left ventricular ejection fraction by echocardiography at 6 months | 6 months
  Evaluating cardiac function using Left ventricular ejection fraction etc. by echocardiography. Assessing change from baseline to 6 months.
Serum free fatty acid levels at 3 months | 3 months
  Analysing concentration of fatty acids in serum using HPLC method. Assessing change from baseline to 3 months.
Serum free fatty acid levels at 6 months | 6 months
  Analysing concentration of fatty acids in serum using HPLC method. Assessing change from baseline to 6 months.

OTHER OUTCOMES:
Incidence, severity, seriousness, causality, and outcomes of adverse events | 6 months
  A frequency counting of the adverse events. LLT code will be assigned to the reported adverse event using the MedDRA dictionary.

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Hirano, MD, Ph.D, Principal Investigator — Department of Cardiovascular Medicine, Faculty of Internal Medicine, Graduate School of Osaka University, Japan; Elena M Pennisi, MD, Ph.D, Principal Investigator — Department of Neurology, San Filippo Neri Hospital, Rome, Italy
Locations (7):
- Italy (4):
  - IRCCS San Raffaele, Rome, Lazio
  - San Filippo Neri Hospital, Rome, Lazio
  - Catholic University, Milan, Lombardy
  - Fondazione Ospedale San Camillo IRCCS, Lido, Venice
- Japan (3):
  - Aomori Prefectural Chuo Hospital, Aomori, Aomori
  - Tohoku University, Sendai, Miyagi
  - Graduate School of Osaka University, Suita, Osaka